CLINICAL TRIAL: NCT00485914
Title: Worksite Vocational Rehabilitation Intervention to Improve Employment Outcomes for Persons With Arthritis?
Brief Title: Work Interventions to Improve Employment Outcomes for Persons With Rheumatoid Arthritis and Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H133B031120-Project 3
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
Keywords: employment; work
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-site work evaluation (Experimental): Participants will receive one-to-one contact with an occupational therapist and an individualized work plan
  Interventions: Behavioral: On-site work evaluation
- Educational material (Active Comparator): Participants will receive educational materials to develop strategies to compensate for limitations caused by their condition
  Interventions: Behavioral: Educational material

INTERVENTIONS:
Behavioral: On-site work evaluation — Researchers will measure the effects of worksite assessment through an on-site work evaluation by an occupational therapist on a person's job satisfaction, capacity to perform work duties, income, health status, and psychological well-being. The scope of the information will be through one-to-one contact and an individualized work plan. The strategies will include recommendations for work behaviors, ergonomic and body mechanics considerations, and modifications for job tasks, equipment, and space.
  Arms: On-site work evaluation
Behavioral: Educational material — Researchers will measure the effects of worksite assessment through educational materials on a person's job satisfaction, capacity to perform work duties, income, health status, and psychological well-being. The scope of the information will be through educational materials to develop strategies to compensate. The strategies will include recommendations for work behaviors, ergonomic and body mechanics considerations, and modifications for job tasks, equipment, and space.
  Arms: Educational material

SUMMARY:
To determine if worksite based functional evaluation/intervention provided by occupational therapists improves employment outcomes for persons with arthritis.

DETAILED DESCRIPTION:
Arthritis is second only to heart disease as a cause of work-related disability with significant financial costs associated with the loss of work for persons with arthritis. Many persons with arthritis have physical impairments which affect their ability to work, with 50% of persons with rheumatoid arthritis leaving employment within 10 years of diagnosis. Risk factors predicting employability, length of employment and worksite accommodations for workers with arthritis have been well documented. Variables predicting work cessation include blue collar jobs and more physically demanding jobs, an older age of the worker, lower education, perceived job strain, social support of co-workers and supervisors, job satisfaction, and self-efficacy. Recent studies of self-report by persons with arthritis identified the use of worksite accommodations such as others providing assistance at work, job autonomy, time flexibility, and use of special equipment. Unknown is the effect of on-site work interventions. The need exists to determine if the provision of strategies for physical accommodations, worksite modifications, and assistive technologies at the individual's job site improves the ability of persons with arthritis to continue working.

This is a randomized clinical trial to investigate the efficacy of a worksite based intervention to improve the employment outcomes of persons with rheumatoid (RA) or osteoarthritis (OA). Persons with RA or OA who have arthritis related work difficulties will have an occupational therapist provide a worksite evaluation and subsequent training in strategies to accommodate arthritis related physical impairments and improve job performance and satisfaction. Participants in control group will be provided with educational printed materials related for a self-initiated worksite evaluation of musculoskeletal and environmental risks at the worksite for persons with arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis or osteoarthritis diagnosed by a rheumatologist
* Competitively employed; full or part time
* Reporting arthritis-related employment difficulties
* Agree to participate in a work site evaluation

Exclusion Criteria:

* Systemic complications of RA (e.g., vasculitis)
* Organic Brain Syndrome
* Uncontrolled psychiatric disorders
* Uncontrolled medical conditions (e.g., active cancer)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2003-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Arthritis Impact Measurement Scale-2, Brief Symptom Inventory, Job Satisfaction Survey, Occupational Data information, Work History, Employment Status, Financial Information | Scores at baseline, 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: George Johnstone, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No